CLINICAL TRIAL: NCT00430690
Title: Acoustic Startle Reduction In Cocaine Dependence
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erica Duncan, MD, Associate Professor, Emory University
Other Study IDs: IRB00002489; R01DA018294-01A2 (NIH)
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and extracted DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Cocaine dependent subjects
  Interventions: Procedure: acoustic startle testing
- 2: Healthy controls
  Interventions: Procedure: acoustic startle testing
- 3: Siblings of cocaine dependent subjects
  Interventions: Procedure: acoustic startle testing

INTERVENTIONS:
Procedure: acoustic startle testing — acoustic startle testing: listening to sounds through headphones while the eyeblink component of the acoustic startle reflex is recorded with small surface electrodes

SUMMARY:
Chronic cocaine administration leads to changes in brain function that persist long after the acute withdrawal phase. The acoustic startle response (ASR) is a well characterized reflexive response to a sudden acoustic stimulus. The ASR is mediated by a simple 3-synapse subcortical circuit; it is modulated in part by brain areas and neurotransmitters associated with cocaine administration. Our initial study and subsequent replication reveals a profound diminution of the ASR in cocaine-dependent subjects after a brief period of abstinence. Our preliminary findings indicate that first degree relatives of cocaine-dependent subjects also have reduced startle compared to healthy controls. The findings of low ASR in rats and humans during cocaine washout and low ASR in family members suggests there may be both a trait and state component of the startle reductions we have reported.

The central objectives of this proposal are to dissect this finding with regard to its development and persistence in early and later phases of cocaine abstinence in humans; to ascertain whether startle reduction and its potential normalization during later abstinence is a predictor of clinical course in human subjects with cocaine dependence; and to examine whether startle reduction is, at least in part, a vulnerability trait for the development of cocaine dependence. This latter Aim will be carried out in humans by testing siblings of cocaine-dependent subjects.

Cocaine dependence is an enormous public health problem. The significance of this work lies in the potential for the ASR reduction to serve as a reliable, easily repeatable biological measure of cocaine-induced brain changes that may enhance outcome prediction so that tailored treatments may be directed at those patients most vulnerable to relapse, given the restriction of resources for available for substance abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

Cocaine dependent subjects:

1. males or females,
2. age 18-80,
3. with a DSM-IV diagnosis of cocaine dependence,
4. a usage history characterized by a minimum of 1 year of at least $50 per day or weekly binges of at least $200 of cocaine use.

Exclusion Criteria:

1. current clinically significant medical illness (including HIV, because of possible confound of neurological involvement),
2. current or past neurological illness, and no history of head trauma with loss of consciousness ≥ 5 minutes because of the possible confound of neurological damage to startle-modulating brain areas,
3. other Axis I psychiatric disorder currently or in the previous three months with the exception of substance induced disorders as determined by SCID,
4. history of schizophrenia, schizoaffective disorder, posttraumatic stress disorder, or bipolar disorder,
5. known hearing impairments (intact hearing will be insured by brief audiology screening),
6. dependence on other drugs or alcohol within the previous 6 months, as confirmed by ASI.

Healthy controls:

1. males or females,
2. age 18-80.

Exclusion criteria:

1. history of any Axis I psychiatric illness or history of treatment as determined by SCID Axis I,
2. substance dependence or abuse history by ASI and SCID,
3. no current clinically significant medical illness (including HIV),
4. current or past neurological illness, or history of head trauma with loss of consciousness ≥ 5 minutes because of the possible confound of neurological damage to startle-modulating brain areas,
5. known hearing impairments (intact hearing will be insured by brief audiology screening),
6. Axis I disorder, including substance dependence, in first degree family member.

Family members of cocaine subjects:

1. males or females,
2. age 18-80,
3. family member of cocaine-dependent subject enrolled in study.

Exclusion criteria:

1. history of any Axis I psychiatric illness or history of treatment as determined by SCID Axis I,
2. substance dependence history by ASI and SCID, or substance abuse within the prior 5 years,
3. no current clinically significant medical illness (including HIV),
4. current or past neurological illness, or history of head trauma with loss of consciousness,
5. known hearing impairments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with cocaine dependence who are entering substance abuse treatment; siblings of these subjects; and healthy controls
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2011-07-19 (Actual); Study Completion 2011-07-19 (Actual)

PRIMARY OUTCOMES:
Acoustic startle magnitude | at baseline
  Magnitude of acoustic startle response as measured by electromyography of eyeblink.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Duncan, MD, Principal Investigator — Emory University / Atlanta VA
Locations (1):
- Atlanta Veterans Adminstration Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No